CLINICAL TRIAL: NCT07136701
Title: Study in Risk Factors, Prognosis, Clinicopathological and Metabolic Characteristics Between Early- and Late-Onset Pancreatic Neuroendocrine Tumors: A Multicenter Retrospective Study
Brief Title: Risk Factors, Prognosis, Clinicopathological and Metabolic Characteristics of EO- vs LO-PanNETs
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: China-Japan Friendship Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Hanxiang Zhan, Chief Physician, Department of Pancreatic Surgery, Qilu Hospital of Shandong University
Other Study IDs: KYLL-2025-07-004
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Neuroendocine Neoplasms (pNETs)
Keywords: EO-PanNET

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Early-onset pancreatic neuroendocrine tumors group: This group comprises patients diagnosed with pancreatic neuroendocrine tumors before the age of 50 years. All cases were histopathologically confirmed and treated at one of the participating centers.
- Late-onset pancreatic neuroendocrine tumors group: This group comprises patients diagnosed with pancreatic neuroendocrine tumors at or after the age of 50 years. All cases were histopathologically confirmed and treated at one of the participating centers.

SUMMARY:
The aim of this observational multicenter retrospective cohort study is to evaluate the differences in risk factors, prognosis, clinicopathological and metabolic characteristics between early-onset pancreatic neuroendocrine tumors (EO-PanNETs) and late-onset pancreatic neuroendocrine tumors (LO-PanNETs).

The main questions it aims to answer are:

Are there distinct clinical, pathological, and metabolic profiles in EO-PanNETs compared with LO-PanNETs? Do EO-PanNETs have different prognostic outcomes compared with LO-PanNETs? Researchers will compare EO-PanNET patients with LO-PanNET patients and with matched nonmalignant controls to assess differences in tumor characteristics and associated metabolic conditions.

Participants will:

Provide retrospective clinical, pathological, and metabolic data from hospital records.

Have survival and recurrence outcomes assessed through follow-up data review.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older; histopathologically confirmed pancreatic neuroendocrine tumor by surgical resection or biopsy.

Exclusion Criteria:

* Pancreatic neuroendocrine carcinoma; incomplete pathological data; received antitumor treatment prior to presentation; with other malignanies or malignant history.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised adult patients (≥18 years) diagnosed with pancreatic neuroendocrine tumors (PanNETs) between 2013 and 2024. All cases had a histopathologically confirmed diagnosis and received treatment at one of the participating centers. Patients were excluded if they had poorly differentiated neuroendocrine carcinoma, mixed neuroendocrine-non-neuroendocrine neoplasm, undefined tumor differentiation, recurrent disease, non-initial treatment, or a history of other malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause or the date of the last follow-up, whichever came first, assessed up to 12 years

SECONDARY OUTCOMES:
Disease-specific survival | From date of diagnosis until death due to PanNETs, up to 12 years
Progression-free survival | From date of diagnosis until the date of disease recurrence or death from any cause, whichever came first, assessed up to 12 years.
Disease-free survival | From date of surgery until first documented recurrence, metastasis, or death from any cause, assessed up to 12 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR